CLINICAL TRIAL: NCT01030874
Title: Effect of Treatment of Orthostatic Hypotension on a Rehabilitation Unit
Brief Title: Orthostatic Hypotension Treatment on Rehab Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: E7278-R
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Orthostatic Hypotension; Falls
Keywords: hypotension, orthostatic; falls; rehabilitation; blood pressure; aging
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Medication Review; Educational Status; Exercise; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Rehabilitation Care (No Intervention): Usual rehab care
- Experimental Treatment/Medication Review (Experimental): Treatment for, and prevention of, orthostatic hypotension
  Interventions: Other: Medication review; Other: Nutrition/Salt intake; Other: Education; Other: Exercise; Other: Drug Recommendations

INTERVENTIONS:
Other: Medication review — Current scheduled and as needed medications will be reviewed. Those medications with potentially hypotensive actions will be identified. There will be a joint review by Provider, Pharmacist, and Research staff of those medications and the patient's current clinical status. Plan to continue, decrease, discontinue, or substitute will be made. Examples include substitution of tamsulosin for prazosin in treating benign prostatic hypertrophy, reduction of furosemide dose for patient with stable congestive heart failure, change of sleeping medication from trazodone to lorazepam or zolpidem; change of antidepressant therapy or neuroleptic therapy to one with less hypotensive effects.(Mader 1989); (Poon and Braun 2005);(Mader 2006); (2008).
  Other Names: Chart review
  Arms: Experimental Treatment/Medication Review
Other: Nutrition/Salt intake — Current diet orders and meal consumption will be reviewed for sodium and fluid intake. Liberalization of calories, fluid, addition of salt packets to tray, or addition of salty foods/beverages (V8) will be considered as appropriate. Subjects receiving tube feedings will have water flushes replaced with saline flushes. Subjects with a history of congestive heart failure will be liberalized slowly and monitored closely by both the research and treatment team.
  Other Names: Review orders; Change nutrition/Salt intake orders
  Arms: Experimental Treatment/Medication Review
Other: Education — The research intervention staff will review symptoms of OH with patient/family and explain pathophysiology using a standardized pt information handout (NINDS 2007), subjects will be encouraged to spend maximal time out of bed, and to ambulate on ward as much as possible.
  Arms: Experimental Treatment/Medication Review
Other: Exercise — The patient's PT and/or Provider will review patient function for the ability to perform appropriate exercises and train patients (Ten Harkel, van Lieshout et al. 1994); (Bouvette, McPhee et al. 1996). Research staff will reinforce using these exercises while standing.
  Other Names: Physical therapy
  Arms: Experimental Treatment/Medication Review
Other: Drug Recommendations — The protocol permits the study physician to recommend medications for orthostatic hypotension. The patient's clinical team can implement, ignore, or modify these recommendations and only the clinical team can write orders for them. Fludrocortisone may be given 0.05mg at bedtime up to 0.2mg twice a day (Ten Harkel, Van Lieshout et al. 1992). Subjects with a history of congestive heart failure or peripheral edema will be carefully monitored. Sodium chloride tablets may be given starting at 1gm daily and increased to 2 gms twice daily [Mukai 2002; Grubb 2003]. Subjects with a history of congestive heart failure or peripheral edema will be carefully reviewed and monitored closely by the research staff and the treatment team. Midodrine may be given 2.5-5mg daily to three times daily [Low, 1997]. The dose will be started at 2.5mg every morning and then increased to 5mg every morning, then 5mg every morning and afternoon, then 5mg three times a day.
  Other Names: Consultant recommendation
  Arms: Experimental Treatment/Medication Review

SUMMARY:
For patients recovering from acute illness, the ability to stand, walk, climb stairs, and participate in therapy are critical to their recovery and eventual discharge to the least restrictive environment. Orthostatic hypotension is a common finding in medically ill adult and elderly patients and is a potentially reversible contributor to functional impairment. This 4-year project will be a randomized controlled trial of a multidisciplinary-multicomponent intervention to determine whether routine identification and treatment of OH improves functional outcomes such as: balance, fall rates, therapy participation, length of stay, transfer to acute care hospital, and discharge location. Routine screening and management of OH may improve outcomes for rehabilitation and long term care patients, as well other high-risk patient populations.

DETAILED DESCRIPTION:
Objectives Orthostatic hypotension (OH) is a condition that contributes to falls, dizziness, syncope, transient ischemic attack, and impaired functional status. OH is defined specifically as a 20mmHg drop in systolic, and/or a 10mmHg drop in diastolic BP within 3 min of standing. The objectives of this study are to: (1) Examine the effect of OH treatment on functional outcomes, and OH prevalence during a subject's inpatient stay, and (2) Evaluate whether OH treatment during a subject's inpatient stay affects fall prevalence, and functional outcomes by 12 months after discharge.

Plan This 4-year project will be a randomized controlled trial of a multidisciplinary-multicomponent intervention to improve OH in patients admitted to Nursing Home (NH) and rehabilitation settings. During the 37-month enrollment period, the investigators expect to consent 350 subjects who will be randomized into intervention and control groups (175 subjects each). During their stay, subjects in the intervention group will receive a standardized treatment for their OH, or to prevent OH, while those in the control group will receive usual care. The investigators expect that 85% will remain in the study until they are discharged from the NH/rehabilitation unit. Following discharge, the investigators will conduct weekly phone calls to monitor incidence of falls for one month. Subsequently, at 12-months post-discharge, the investigators will conduct a chart review, and the study will terminate. The investigators expect 85% of the subjects discharged from the NH/rehabilitation unit that were enrolled in the study will remain in the study at 12-months post discharge. The investigators performed a "pilot" study on up to 10 subjects while waiting for adequate staffing to conduct the study with blinded data collectors.

Methods The investigators will evaluate OH blood pressure responses, symptoms during standing, and whether there are any specific adverse outcomes related to treatment. In addition, the investigators will evaluate whether treatment of OH improves: motor functional independence measure (mFIM) scores, therapy participation, length of stay, transfer to the acute care hospital, discharge location, and mortality.

Clinical Relevance OH is a very common finding in many medically ill adult and elderly patients, and is associated with falls, syncope, and hip fractures. More aggressive screening (possibly the 6th vital sign) and management of this condition may improve outcomes for rehabilitation and long term care patients at the investigators' site as well other high-risk patient populations.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the nursing home, and rehabilitation unit

Exclusion Criteria:

* hospice admission
* respite admission
* long-stay admission
* transplant admission
* inability to stand
* expected length of stay less than 14 days
* patients specifically admitted for treatment of OH
* cognitive dysfunction of such a severity that the admitting provider does not feel the patient could understand the study and safely participate in the data collection
* administrative exclusion, such as safety concerns of staff due to violent tendencies of patient

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2011-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Helfand, MD MPH MS, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1/ Inpatient Rehabilitation Care (Usual Care): Usual rehab care
- Arm 2 / Treatment for, and Prevention of, Orthostatic Hypotension.: Orthostatic hypotension interventions
Period: Overall Study
Arm/Group | Arm 1/ Inpatient Rehabilitation Care (Usual Care) | Arm 2 / Treatment for, and Prevention of, Orthostatic Hypotension.
Started | 178 (1 with impaired decision making capacity) | 178 (1 with impaired decision making capacity)
Completed | 160 | 162
Not Completed | 18 | 16
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Discharged in first 2 weeks | 17 | 16

BASELINE CHARACTERISTICS:
Population: Excluding one participant that withdrew and did not want data to be included.
Groups:
- Arm 1: Usual rehab care
- Arm 2: Treatment for, and prevention of, orthostatic hypotension
  Medications will be reviewed to identify those with potentially hypotensive actions. After joint review by Provider, Pharmacist, and Research staff, a plan to continue, decrease, discontinue, or substitute will be made. Examples include substitution of tamsulosin for prazosin in treating benign prostatic hypertrophy, reduction of furosemide dose for patient with stable congestive heart failure, change of sleeping medication from trazodone to lorazepam or zolpidem; change of antidepressant therapy or neuroleptic therapy to one with less hypotensive effects.(Mader 1989); (Poon and Braun 2005);(Mader 2006); (2008).
  Nutrition/Salt intake: Current diet orders and meal consumption will be reviewed for sodium and fluid intake. Liberalization of calories, fluid, addition of salt packets to t
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 177 | 178 | 355
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (10.5) | 65.0 (11.7) | 66.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 164 | 168 | 332
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 156 | 163 | 319
  Unknown or Not Reported | 18 | 11 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 8 | 5 | 13
  White | 143 | 151 | 294
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 18 | 18 | 36
Education [Mean (Standard Deviation); unit: years] | 13.6 (2.3) | 13.6 (2.5) | 13.6 (2.4)
Smoker [Count of Participants; unit: Participants]
  Never | 32 | 34 | 66
  Current | 42 | 54 | 96
  Former | 98 | 84 | 182
  Missing | 5 | 6 | 11
Location Admitted From [Count of Participants; unit: Participants]
  VA Hospital | 114 | 116 | 230
  Home | 29 | 32 | 61
  Nursing Home | 8 | 5 | 13
  Homeless | 1 | 0 | 1
  Outside Hospital | 23 | 22 | 45
  Other | 2 | 3 | 5
Falls in past month [Count of Participants; unit: Participants]
  Yes | 55 | 59 | 114
  No | 113 | 112 | 225
  Missing | 9 | 7 | 16
Falls in past year [Median (Full Range); unit: Falls] | 1 [0 to 40] | 1 [0 to 60] | 1 [0 to 60]

OUTCOME MEASURES:

1. Primary Outcome: Orthostatic Hypotension at Discharge
Description: Patients were categorized as having orthostatic hypotension at discharge if they had a decrease in systolic BP > 30 or diastolic pressure >15 mm Hg at 1 or 3 minutes after standing compared with the mean of the supine values, on two or more readings in the last week of admission.
Time Frame: Duration in rehabilitation facility (time to discharge or transfer) varied for participants. For patients included in the analysis, mean length of stay was 41.2 days (median 31 days), with a range of 10 to 90 days.
Population: Analyses were restricted to patients for which OH status could be determined at both baseline and discharge. This required at least four blood pressure assessments, with at least two assessments each in separate weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 2: Treatment for, and prevention of, orthostatic hypotension
  Medication review: Current scheduled and as needed medications will be reviewed. Those medications with potentially hypotensive actions will be identified. There will be a joint review by Provider, Pharmacist, and Research staff of those medications and the patient's current clinical status. Plan to continue, decrease, discontinue, or substitute will be made. Examples include substitution of tamsulosin for prazosin in treating benign prostatic hypertrophy, reduction of furosemide dose for patient with stable congestive heart failure, change of sleeping medication from trazodone to lorazepam or zolpidem; change of antidepressant therapy or neuroleptic therapy to one with less hypotensive effects.(Mader 1989); (Poon and Braun 2005);(Mader 2006); (2008).
  Nutrition/Salt intake: Current diet orders and meal consumption will be reviewed for sodium and fluid intake. Liberalization of calories, fluid, addition of salt packets to t
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 151 | 150
Participants | 39 | 44
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Other; p = 0.6, Regression, Logistic; Adjusted for whether patient had orthostatic hypotension at baseline; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.67 to 1.99] — Arm 2 is in the numerator of OR calculation

2. Secondary Outcome: Falls 30 Days After Discharge
Description: Falls 30 days after discharge was dichotomized to indicate whether a patient had at least one fall during the 30 days after discharge versus no falls.
Time Frame: Time to discharge varied for participants. For patients included in the analysis, mean length of stay was 41.2 days (median 31 days), with a range of 10 to 90 days, so 30 days after discharge ranged from 40 days to 120 days.
Population: Analysis restricted to patients with post-discharge falls data.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 161 | 159
Participants | 18 | 20
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Other; p = 0.3, Regression, Logistic; Adjusted for whether patient had orthostatic hypotension at discharge; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.74 to 3.24] — Arm 2 is in the numerator of OR calculation

ADVERSE EVENTS:
Time Frame: Inpatient all-cause mortality was collected ("inpatient" means while in inpatient rehabilitation or in an acute care hospital after transfer from inpatient rehabilitation.) Transfers to an acute care hospital from the rehabilitation facility were also measured. Duration in rehabilitation facility varied for participants included in the analyses (range 10-90 days, median 31 days, mean 41.2 days).
Description: "Other (Not Including Serious) Adverse Events" were not measured and the following fields are not applicable:
  1. "Frequency Threshold for Reporting Other (Not Including Serious) Adverse Events"
  2. "Total Number Affected by Any Other (Not Including Serious) Adverse Event Above the Frequency Threshold"
  Because "not applicable" is not an option, we entered zero values in these fields, indicating they were not relevant and were not measured.
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 13/177 | 14/178
Serious Adverse Events (participants affected / at risk) | 22/177 | 26/178
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=177) | Arm 2 (N=178)
Hospitalization (General disorders) | 22 | 26 — This refers to hospitalization in an acute care facility for any reason. Reasons for transfer could include exacerbation of a comorbid condition or an emergent condition.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=0) | Arm 2 (N=0)
Other (Not Including Serious) Adverse Events (General disorders) | 0 (0) | 0 (0) — Other (Not Including Serious) Adverse Events were not measured or recorded. The threshold for recording was hospitalization or death.

LIMITATIONS AND CAVEATS:
In 2013 a new PI was appointed. The protocol, practices, and procedures for the study were reviewed, and collection of some data items was discontinued because of measurement problems or a high rate of missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes